CLINICAL TRIAL: NCT07053956
Title: Impact of Chewing Gum on FeNO Levels in Patients With Bronchial Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Jens Spießhöfer, MD, PhD, RWTH Aachen University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 24-515
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Asthma Bronchiale; FeNO; Chewing Gum
Keywords: Asthma bronchiale; FeNO; Chewing Gum
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: Single-center interventional randomized case-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chewing gum arm (Active Comparator): Patients admitted to our outpatient clinic for bronchial asthma undergo regular FeNO measurements. If the value is ≥ 25 ppb (elevated), the patients are randomized into two groups after obtaining their consent. In the control group, a FeNO measurement is performed again after 15 minutes. In the second group, the FeNO measurement is measured again after 15 minutes of consuming sugar-free, antioxidant-containing chewing gum. The following data are then collected and documented from the patients: age, gender, height, weight, smoking status, current medication, other illnesses, whole body lung function test, and laboratory tests (eosinophils, IgE). Participation in the study will not change the course of the patient's stay in our clinic.
  Interventions: Other: Chewing Gum
- Control arm (Sham Comparator): Patients admitted to our outpatient clinic for bronchial asthma undergo regular FeNO measurements. If the value is ≥ 25 ppb (elevated), the patients are randomized into two groups after obtaining their consent. In the control group, a FeNO measurement is performed again after 15 minutes. In the second group, the FeNO measurement is measured again after 15 minutes of consuming sugar-free, antioxidant-containing chewing gum. The following data are then collected and documented from the patients: age, gender, height, weight, smoking status, current medication, other illnesses, whole body lung function test, and laboratory tests (eosinophils, IgE). Participation in the study will not change the course of the patient's stay in our clinic.
  Interventions: Other: Chewing Gum

INTERVENTIONS:
Other: Chewing Gum — Patients admitted to our outpatient clinic for bronchial asthma undergo regular FeNO measurements. If the value is ≥ 25 ppb (elevated), the patients are randomized into two groups after obtaining their consent. In the control group, a FeNO measurement is performed again after 15 minutes. In the second group, the FeNO measurement is measured again after 15 minutes of consuming sugar-free, antioxidant-containing chewing gum. The following data are then collected and documented from the patients: age, gender, height, weight, smoking status, current medication, other illnesses, whole body lung function test, and laboratory tests (eosinophils, IgE). Participation in the study will not change the course of the patient's stay in our clinic.

SUMMARY:
The aim of the study is to investigate the influence of chewing gum consumption on FeNO levels in asthma patients in order to avoid systematic errors in treatment decisions.

DETAILED DESCRIPTION:
FeNO measurement is a non-invasive, available measure both for the diagnostic workup of patients with suspected bronchial asthma and for therapy management after a confirmed diagnosis. In patients with bronchial asthma, FeNO is a biomarker of airway inflammation. The recommended lower FeNO limits of the American Thoracic Society (ATS) are < 25 ppb in adults. A significantly elevated FeNO level (≥ 50 ppb), especially in the presence of increased blood eosinophil counts (≥ 300/µl), indicates an increased risk of exacerbation. Furthermore, patients with elevated FeNO levels are generally (inhalative cortison treatment; ICS) responsive. Conversely, elevated FeNO levels (especially FeNO levels > 50 ppb) during ICS therapy, despite clinical stability, argue against a reduction in the ICS dose.

Elevated FeNO levels during ICS therapy can occur due to poor treatment adherence. However, persistently elevated FeNO levels despite ICS therapy can also indicate inflammation in the airways that does not respond to further increases in the ICS dose. In summary, measuring airway inflammation using FeNO is an important component in the diagnosis and management of asthma.

It is already known that acute tobacco smoke exposure lowers FeNO levels in patients with asthma. Furthermore, FeNO levels are strongly influenced by factors such as infections, stress, or exposure to pollutants. Food containing nitrates (salad, sausage) can increase FeNO levels. Our patients are informed about these known factors so that they can avoid exposure prior to their medical consultation and examination. Conversely, it is suspected that chewing gum, which influences the oral flora, may lower FeNO levels, which would lead to false-negative FeNO levels and thus potentially prevent better diagnosis and treatment of asthma. However, to the best of our knowledge no study has yet examined the influence of chewing gum on FeNO levels.

Hence, the aim of the study is to investigate the influence of chewing gum consumption on FeNO levels in asthma patients in order to avoid systematic errors in treatment decisions.

Patients admitted to our outpatient clinic for bronchial asthma undergo regular FeNO measurements. If the value is ≥ 25 ppb (elevated), the patients are randomized into two groups after obtaining their consent. In the control group, a FeNO measurement is performed again after 15 minutes. In the second group, the FeNO measurement is measured again after 15 minutes of consuming sugar-free, antioxidant-containing chewing gum. The following data are then collected and documented from the patients: age, gender, height, weight, smoking status, current medication, other illnesses, whole body lung function test, and laboratory tests (eosinophils, IgE). Participation in the study will not change the course of the patient's stay in our clinic.

ELIGIBILITY:
Inclusion Criteria:

1. have known bronchial asthma with a FeNO level ≥25 ppb at regular medical checkups
2. are of legal age
3. are mentally and physically capable of understanding the significance and scope of the study and obeying the instructions of study personnel
4. are legally competent and have signed the informed consent form.

Exclusion Criteria:

1. Current or past medically relevant illness or treatment that could impact the evaluability of the study.
2. FeNO levels < 25 ppb
3. Medical contraindications to conducting FeNO measurements
4. Expected unwillingness to actively participate in study-related measures.
5. Known allergies or intolerances to the contents of chewing gum
6. Smoking, alcohol consumption, mouthwash use, chewing gum/candy/lettuce/spinach/kale/beetroot/radish/sausage consumption, or exercise on the day of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
FeNO measurement after 15 minutes of consuming sugar-free, antioxidant-containing chewing gum | 15 Minutes
  FeNO measurement is measured again after 15 minutes of consuming sugar-free, antioxidant-containing chewing gum

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Maria Aetou Aetou, Principal Investigator — RWTH Aachen University Hospital; Professor Michael Dreher Dreher, Study Director — RWTH Aachen University Hospital
Locations (2):
- Germany (2):
  - University Hospital Aachen, Aachen, Aachen
  - Department of Pneumology and Intensive Care Medicine, RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request study protocol and SAP and data will be shared in pseudonomyzed form
Supporting Information: Study Protocol, SAP
Time Frame: Until further notice